CLINICAL TRIAL: NCT01395225
Title: Standardising an Approach for Analysis of Lymph Node Specimens From Radical Cystectomy With Pelvic Lymph Node Dissection Through the Use of an Organic Fat-emulsifying Agent
Brief Title: Lymph Node Processing Protocol for Radical Cystectomy and Pelvic Lymph Node Dissection in Bladder Cancer
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Urologic Oncology Group (Other)
Responsible Party: Sponsor
Other Study IDs: H11-00748
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Bladder Cancer; Transitional Cell Carcinoma
Keywords: Fat Emulsifying; Radical Cystectomy; Pelvic Lymph Node Dissection; Pathological Lymph Node Processing; Bladder Cancer; Transitional Cell Carcinoma; Urothelial Cell Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All Patients: There will be no separate cohorts in this study. All patients will have their specimens processed by conventional means and by the study method. The conventional means will be the control for the study method.

SUMMARY:
When the bladder is removed for bladder cancer, pelvic lymph nodes (LN) are also removed. While the anatomic extent of this LN dissection is critical, the investigators often use the number of LN removed as a measure of the extent, which in turn is essential for determining the patient's further treatment and prognosis. The LN count, however, is also dependent on the pathologist's processing of the LN tissue, and the standards for this processing are poorly defined. The goal of this study is to establish a standardized method for processing and analyzing lymph node specimens. The investigators hypothesize that if an organic solvent is used to remove excess fat from the lymph nodes that the investigators will discover more clinically significant nodes in a more reproducible fashion when compared to the current method.

DETAILED DESCRIPTION:
PURPOSE:

This research aims to compare the clinical significance of the use of a fat emulsifying protocol versus the current standard in the processing of lymph node specimens following radical cystectomy and pelvic lymph node dissection.

HYPOTHESIS:

The investigators hypothesize that the use of a fat-emulsifying protocol in the processing of lymph nodes harvested at the time of radical cystectomy will increase the proportion of patients found to have lymph node metastases when compared to the current standard technique.

JUSTIFICATION:

The mainstay of management of muscle invasive bladder cancer is radical cystectomy with pelvic lymph node dissection (PLND). Despite optimal multimodal therapy, approximately half of patients with invasive bladder cancer die of their disease. Efforts to improve patient outcome have focussed on two principle factors: the delivery of pre-operative chemotherapy and the adequacy of PLND. While a PLND is ultimately defined by its anatomic extent, a popular surrogate measure of extent is the number of lymph nodes removed. Beyond assessing the adequacy of the PLND in the sense of quality of care, the accurate determination of lymph node involvement is essential for the correct staging of the patient, which is used to guide adjuvant therapy and determine patient prognosis. The processing and analysis of the lymph node specimens is therefore critical in multiple ways.

The current convention at Vancouver General Hospital for specimen handling involves the dissection of the nodal specimen by a laboratory technologist in the pathology lab. Only palpable nodes are processed for sectioning and the remaining fat tissue is discarded. The nodal count is determined by the pathologist when reviewing the slides based on a combination of the macroscopic and microscopic examination. This process is highly subjective, depends on the diligence of the technologist's dissection, and limits the final examination to palpable nodes. In the fat emulsifying technique, all fat is dissolved so that the pathologist can visualize and process all nodes. The investigators believe that this may provide for a more standardized and reproducible method in processing lymph nodes.

A standardized and reproducible method for processing lymph nodes is a prerequisite to any use of lymph node counts as a measure of the quality of the PLND. And, it is necessary to allow the comparison of results between centers. Furthermore, standardized methodology is essential to ensure adequate sampling of lymph nodes for clinical staging and prognostication.

OBJECTIVES:

The investigators have designed a prospective trial to compare our current protocol for processing pelvic lymph nodes from radical cystectomy with PLND to a fat-emulsifying protocol. The investigators aim to answer three questions with this trial:

i. While the fat-emulsifying technique will almost certainly identify more nodes than the current technique of manual dissection, and will likely identify more nodal metastases, the aim of this study is to determine whether a more careful analysis will find a greater proportion of patients to have lymph node metastases. This will translate into better staging and prognostication.

ii. The current technique likely misses particularly small lymph nodes that are not easily palpated. The investigators hypothesize that there is no threshold lymph node size below which the risk of metastasis is negligible, and that identification of these smaller nodes is therefore clinically meaningful.

iii. The investigators hypothesize that a fat-emulsifying protocol will remove much of the variability due to human element of manual dissection by the prosector. While the investigators will not test this hypothesis directly, the investigators believe the methodology and photographic documentation of the results will reflect a degree of objectivity in this methodology that is not seen with other techniques.

The ultimate goal of this research proposal is to develop a standardized and reproducible technique that can be used everywhere in order to enhance the care of our patients with invasive bladder cancer.

RESEARCH METHOD:

Patients:

All patients who undergo radical cystectomy with pelvic lymph node dissection at Vancouver General Hospital (VGH) will be invited to participate in this prospective study. Patients with clinical stage T1-4,N0,M0 bladder cancer will be invited to participate in the study and will be enrolled after informed consent is obtained.

Surgical technique:

The extent of lymph node dissection will be defined as either conventional (up to bifurcation of common iliac artery) or extended (at least up to the aortic bifurcation) and will be determined by the surgeon on a case-by-case basis. Dissection of the pre-sacral lymph nodes is also up to the surgeon. Objective documentation of the extent of node dissection will be assured by intra-operative photography in every case.

Pathologic processing of PLND specimen:

Each specimen will be analyzed by both conventional means and by a fat-emulsifying protocol. The current convention at Vancouver General Hospital for specimen handling is described above. In this study the pathologist will count the number of nodes dissected by the prosector according to this current protocol. The tissue remaining after removal of the grossly palpable lymph nodes will be submitted for processing by the fat-emulsifying protocol, which is identical to the LNRS ("lymph node removing solution") protocol defined by Koren et al. This consists of placement of the entire specimen in a specialized solution for 12 hours. The solution is a mixture of 95% ethanol, diethyl ether, glacial acetic acid and buffered formalin in a ratio by volume of 6.5:2:0.5:1 Specimens so treated will be photographed for objective documentation of the nodal count. The additional nodes are then embedded in paraffin, sectioned at 2 mm intervals, and stained with eosin and hematoxylin. The total number of nodes, their size and presence of metastasis will be recorded.

Data collection:

Demographic, clinical and pathological information will be recorded prospectively. Demographic variables analyzed will include: age, sex, weight, height and race. Clinical variables will include: date of cancer diagnosis, clinical and pathologic stage at diagnosis and at time of surgery (TNM staging), date of radical cystectomy, history of intravesical chemotherapy, other medical co-morbidities and prior abdominal surgeries, extent of lymph node dissection, and complications during the procedure. Pathological variables will be recorded for the findings on both the conventional and fat-emulsifying protocols. The number, size and presence of metastasis for each node found will be recorded.

STATISTICAL ANALYSIS:

Outcome measure:

The primary outcome will be the proportion of patients found to have lymph nodes metastases on pathologic examination. Specifically, the difference in proportion of specimens found to contain nodal metastases using the fat-emulsifying protocol compared to the conventional lymph node processing will be analyzed. Secondary outcome measures will be: the total number of lymph nodes and the total number of lymph node metastases counted by both techniques and the relationship between the size of lymph node and the presence of metastatic carcinoma.

Sample size calculation:

An increase in the identification of nodal metastases by 15% (fat-emulsifying compared to conventional processing) will be considered clinically significant. The current rate of node positivity at the time of radical cystectomy with PLND at VGH is 28%, so that an increase to 43% would be deemed clinically relevant. To detect this difference with a power (1-β) of 80% and an α error of 10%, 125 patients will need be enrolled in each arm of the study.

Analysis of Data:

Data will be analyzed using SPSS software. The independent samples t-test will be used to compare the results from the lymph node analysis when processed by conventional means versus the same nodes processed using the fat-emulsifying protocol (p<0.5). The relationship of size to presence of metastatic disease will be done by linear regression model (p<0.5). A significant difference between the groups will be defined as p<0.05. A biostatistician (Robert Bell) at the Vancouver Prostate Centre will assist with data analysis.

SUMMARY

The investigators have the opportunity with simple and inexpensive technical processing measures to enhance an integral component of our clinical risk stratification in patients with invasive bladder cancer. The investigators can establish a solid foundation in pelvic lymph node counting upon which clinical concepts of lymph node yield and density can be validated. The investigators expect to demonstrate that the fat-emulsifying protocol is easy to adopt, reproducible and suitable for widespread use. It has the potential to impact every patient undergoing radical cystectomy with PLND.

ELIGIBILITY:
Inclusion Criteria:

* All patients who undergo radical cystectomy with lymph node dissection at the Vancouver General Hospital (VGH) for clinical stage T1-4,N0,M0 bladder cancer will be invited to participate in this prospective study.

Exclusion Criteria:

1. Inability to consent to study.
2. Presence of concomitant malignancy.
3. The use of neoadjuvant chemotherapy or radiation therapy.
4. Prior pelvic surgery or radiation that may impair ability to perform adequate pelvic lymph node dissection.
5. If a patient is enrolled but does not undergo a lymph node dissection (for example due to other intraoperative complications), the patient will be excluded from analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who undergo radical cystectomy with lymph node dissection at the Vancouver General Hospital (VGH) for clinical stage T1-4,N0,M0 bladder cancer will be invited to participate in this prospective study.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2011-08; Primary Completion 2013-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with lymph node metastasis on pathologic examination | 2 years
  The primary outcome will be the proportion of patients found to have lymph nodes metastases on pathologic examination. Specifically, the difference in proportion of specimens found to contain nodal metastases using the fat-emulsifying protocol compared to the conventional lymph node processing will be analyzed.

SECONDARY OUTCOMES:
Total number of lymph nodes and lymph node metastasis | 2 years
  Secondary outcome measures will be: the total number of lymph nodes and the total number of lymph node metastases counted by both techniques and the relationship between the size of lymph node and the presence of metastatic carcinoma.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Black, MD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Koren R, Paz A, Lask D, Kyzer S, Klein B, Schwartz A, Gal R. Lymph-node revealing solution: a new method for detecting minute lymph nodes in cystectomy specimens. Br J Urol. 1997 Jul;80(1):40-3. doi: 10.1046/j.1464-410x.1997.00154.x. PMID 9240178